CLINICAL TRIAL: NCT00023543
Title: Reduction of Triglycerides in Women on HRT
Brief Title: Reduction of Triglycerides in Women on Hormone Replacement Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 981; R01HL066468-06 (NIH); R01HL066468 (NIH)
Record Dates: First submitted 2001-09-07; First posted 2001-09-07 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Postmenopause; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Heart Diseases | interventions — Diet, Fat-Restricted; Exercise

ARMS (1):
- 1 (Experimental): Participants will reduce total fat intake to 17 percent of calories, 1300 kilo calories, and increase moderate activity to 150-240 minutes per week to obtain a 10 percent reduction in weight.
  Interventions: Behavioral: Diet, fat-restricted; Behavioral: Exercise

INTERVENTIONS:
Behavioral: Diet, fat-restricted — Reduction in total, saturated, trans fat, cholesterol, calories. Increase in fiber. Promotion of nutrient-dense, high-volume, low calorie foods.
Behavioral: Exercise — Rigorous, stepped care approach to reach 150 min/week of physical activity.

SUMMARY:
The purpose of this study is to test the effect of lifestyle intervention on subclinical cardiovascular disease measures in women taking hormone replacement therapy (HRT).

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular disease is a common cause of morbidity and mortality in older women. Better methods of prevention via health promotion are needed. Estrogen HRT may beneficially affect women's cardiovascular health, based on evidence from observational studies, but recent trial evidence suggests HRT may actually lead to increased risk of cardiovascular disease in new users. Understanding this untoward effect of HRT and how to prevent it is a significant aim.

DESIGN NARRATIVE:

This randomized trial of 500 women on HRT for at least two years, aged 52-60 years, and three or more years postmenopausal will test whether reduction in waist circumference, triglycerides, dense low density lipoprotein cholesterol (LDLc), number of LDL particles, C-reactive protein, and plasminogen activator inhibitor-I (PAI-I) by aggressive diet and exercise, versus a health education control, and will decrease progression or result in regression of measures of subclinical vascular disease. The intervention is designed to reduce total fat intake to 17 percent of calories, 1300 kilo calories, and increase moderate activity to 150-240 minutes per week to obtain a 10 percent reduction in weight. The primary endpoint will be a 20 percent or at least a 20 mg decrease in triglyceride levels, a 5 cm decrease in waist circumference, and a 10 percent decrease in LDLc. This will result in changes in subclinical measurements, including carotid ultrasound, electron beam computer tomography of the coronary artery and aorta, pulse wave velocity, endothelial function, and tonometry of the radial artery. Nuclear magnetic resonance spectroscopy of lipoproteins, inflammatory markers, and estrogen metabolites will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* On HRT for at least two years
* Women 52 to 60 years of age
* Three or more years postmenopausal
* Waist circumference greater than 80 cm
* LDLc between 100 and 160 mg/dl
* Body mass index 25-39.9 kg/m2
* Blood Pressure less than 160/95 mm Hg
* Beck Depression Inventory Score less than 20

Exclusion Criteria:

* Current use of cholesterol-lowering medication
* Diagnosis of diabetes
* On diabetes medication

Ages: 52 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 508 (Actual)
Dates: Start 2001-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Measures of subclinical disease | 5 years
Change in coronary calcium (EBCT) | 5 years
Change in carotid intima media wall thickness | 5 years
Change in vascular stiffness (PWV) | 5 years

SECONDARY OUTCOMES:
Change in waist circumference and weight | 5 years
Change in LDL particles, triglycerides and small, medium and large LDL particles | 5 years
Change in HDL particles | 5 years
Change in insulin and glucose | 5 years
Change in systolic blood pressure, diastolic blood pressure | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lewis H. Kuller, MD, DPH, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Kuller LH, Kinzel LS, Pettee KK, Kriska AM, Simkin-Silverman LR, Conroy MB, Averbach F, Pappert WS, Johnson BD. Lifestyle intervention and coronary heart disease risk factor changes over 18 months in postmenopausal women: the Women On the Move through Activity and Nutrition (WOMAN study) clinical trial. J Womens Health (Larchmt). 2006 Oct;15(8):962-74. doi: 10.1089/jwh.2006.15.962. PMID 17087620
- [Derived] Kuller LH, Pettee Gabriel KK, Kinzel LS, Underwood DA, Conroy MB, Chang Y, Mackey RH, Edmundowicz D, Tyrrell KS, Buhari AM, Kriska AM. The Women on the Move Through Activity and Nutrition (WOMAN) study: final 48-month results. Obesity (Silver Spring). 2012 Mar;20(3):636-43. doi: 10.1038/oby.2011.80. Epub 2011 Apr 14. PMID 21494228
- [Derived] Gabriel KP, McClain JJ, Schmid KK, Storti KL, High RR, Underwood DA, Kuller LH, Kriska AM. Issues in accelerometer methodology: the role of epoch length on estimates of physical activity and relationships with health outcomes in overweight, post-menopausal women. Int J Behav Nutr Phys Act. 2010 Jun 15;7:53. doi: 10.1186/1479-5868-7-53. PMID 20550691